CLINICAL TRIAL: NCT01925391
Title: The Measurement of Intraocular Pressure in Nonglaucomatous Children Under Nitrous Oxide/02/Topical Anesthesia and Sevoflurane/Nitrous Oxide/Topical Anesthesia
Brief Title: The Measurement of Intraocular Pressure in Normal Children Under General Anesthesia With and Without Nitrous Oxide and Anesthetic Eye Drops
Acronym: IOP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jacqueline L Tutiven, Assistant professor of Clinical Anesthesia, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20120451
Record Dates: First submitted 2013-08-12; First posted 2013-08-19 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Glaucoma; Intraocular Pressure; Anesthesia
Keywords: Pediatric glaucoma; Intraocular pressure; pediatric glaucoma diagnosis; Volatiles and intraocular pressure; nitrous oxide; Tetracaine
MeSH Terms: conditions — Glaucoma; Hydrophthalmos

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevoflurane, oxygen, intraocular pressure (Active Comparator): Intraocular measurements under induction with Sevoflurane in oxygen
  Interventions: Drug: Tono-pen XL Applanation tonometer + Ocu-film +
- Nitrous oxide/O2/tetracaine (Active Comparator): intraocular pressures in children undergoing inhalation induction with nitrous oxide in oxygen
  Interventions: Drug: Tono-pen XL Applanation tonometer + Ocu-film +

INTERVENTIONS:
Drug: Tono-pen XL Applanation tonometer + Ocu-film +
  Other Names: Tono-pen Applanation tonometer, Reichert Technologies

SUMMARY:
Pediatric glaucoma is a rare but potentially blinding condition where the pressure in the eye is too high. Diagnosis is based on intraocular pressure (IOP) and assessment of the optic nerve, cornea and other structures. Accurate intraocular pressure measurements in young children is often impossible to obtain in an office setting. Children need sedation or general anesthesia to determine IOP. All volatile general anesthetics affect the IOP. Nitrous Oxide, a weak volatile anesthetic, does not affect IOP in healthy adults. Since Nitrous Oxide has shown to be safe and effective in a variety of practice environments, we want to evaluate the use of nitrous oxide in oxygen to obtain IOP measurements in children.

DETAILED DESCRIPTION:
The investigator's intention is to measure the IOP under nitrous oxide in Oxygen followed by measurements under Sevoflurane in a population of children without glaucoma who are already scheduled to undergo general anesthesia for an elective eye surgery. Normally, induction and maintenance of general anesthesia in children includes the addition of volatile anesthetics such as Sevoflurane. The investigators hypothesize that in children, Nitrous oxide will affect IOP from pre-anesthetic baseline minimally. Hence, when sequential IOP measurements are taken in short intervals ( every 30 seconds times 3), there will be minimal changes during the initial nitrous oxide phase of the induction when compared to the subsequent addition of Sevoflurane.

Subject's parents will be consented and if the subject is old enough to understand the procedure, we will have them also sign an assent to the participation of this study.The child will be randomized to either the nitrous oxide in oxygen and Sevoflurane group or the Nitrous oxide in oxygen alone group or Sevoflurane in oxygen group without Nitrous oxide in the inhalational anesthetic mix.

Subjects will be pre-treated with midazolam via oral administration as a dose of 0.5 - 1 mg/kg not to exceed 20 mg total. If they present with an intravenous line, they will be pre-treated with midazolam at 0.05 - 0.1 mg/kg. All patients receiving preoperative sedation will be monitored as per ASA procedural sedation guidelines.

Once the subject is bought into the operating room, all ASA mandatory vital sign monitors will be connected and tetracaine eye drops ( a fast acting topical anesthetic solution) will be placed on the subject's right eye. The rapid clearance of this short acting topical anesthetic reduces any potential risk for systemic toxicity. Once the drops are in,inhalation induction will begin and an initial attempt at measuring IOP will begin when the pediatric anesthesiologist deems the patient is ready clinically.all vital signs and IOP Measurements will be repeated every 30 seconds three times and recorded for data analysis. Once these measurements are recorded, the case will proceed as scheduled and planned.

ELIGIBILITY:
Inclusion Criteria:

* male or female from 1 year of age to less than 18 years of age
* Out-patients scheduled to undergo examination under anesthesia
* out-patients scheduled to undergo eye surgery for strabismus or oculoplastic procedure.
* ASA status I or II
* female patients who have attained menarche must have negative pregnancy tests at screening

Exclusion Criteria:

* patients that have contraindications to the use of nitrous oxide in oxygen
* glaucoma patients
* patients in whom IOP cannot be measured accurately
* latex allergy patients
* patients allergic to aminoesthers

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Measurement of intraocular pressure in nonglaucomatous children under Nitrous oxide/Oxygen/topical anesthesia and Nitrous oxide/Sevoflurane/oxygen/Topical anesthesia. | Up to 40 weeks
  The investigator's intention is to measure IOP in children, who otherwise will be undergoing elective surgery, under nitrous oxide in oxygen and compare those measurements with those going under anesthesia with Sevoflurane in oxygen. The investigators hypothesize that children pre-sedated for surgery,cooperate with topical eye anesthetics and nitrous oxide in oxygen for IOP measurements and results may reflect pre-anesthetic baseline pressures when compared with an induction with Sevoflurane in oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline L tutiven, Md, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Bascom Palmer Eye Hospital, Miami, Florida
  - Bascom Palmer Eye Hospital, Miami, Florida